CLINICAL TRIAL: NCT04670913
Title: A Single-Arm Phase II Trial of Camrelizumab Plus Apatinib for Advanced Non-Squamous NSCLC Previously Treated With First-Line Immunotherapy
Brief Title: Camrelizumab Plus Apatinib for Advanced Non-Squamous NSCLC Previously Treated With First-Line Immunotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Junling Li (Other)
Responsible Party: Sponsor-Investigator, Junling Li, Prof. Junling Li, Chief Physician, Medical Doctor, PhD Tutor, Internal Medicine-Oncology, Chinese Academy of Medical Sciences Cancer Hospital, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2607
Record Dates: First submitted 2020-11-26; First posted 2020-12-17 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Advanced Non Squamous NSCLC
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); anti-angiogenesis; First-Line Immunotherapy
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus Apatinib (Experimental): Camrelizumab, 200mg, q3w, iv and Apatinib, 250mg, qd, po
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — A human anti-PD-1 monoclonal antibody
  Other Names: SHR-1210
Drug: Apatinib — A tyrosine kinase inhibitor selectively targeting VEGFR-2
  Other Names: Apatinibmesylate

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Camrelizumab plus Apatinib in the treatment of advanced non-squamous NSCLC previously treated with first-line immunotherapy

DETAILED DESCRIPTION:
This trial will evaluate the safety and efficacy of Camrelizumab plus Apatinib in participants with advanced non-squamous NSCLC previously treated with first-line immunotherapy. The primary objective of this pilot study is to determine the Camrelizumab plus Apatinib improves progression-free survival (PFS) . All the efficacy and safety are assessed by investigator : 1) response rate (ORR), 2) duration of response(DoR), 3) overall survival(OS), 4) disease control rate (DCR); the safety and quality of life assessment Explore objective is potential biomarker associated with efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed (infomed consent form, ICF).
2. The best response of first-line immunotherapy was SD or above, and PFS was at least 3 months.
3. Male and female aged ≥18 years and ≤75 years.
4. Subjects with histologically or cytologically-documented non-squamous cell NSCLC who present with Stage IIIB/IV disease or recurrent or progressive disease following multimodal therapy.
5. Patients who are unwilling to receive chemotherapy after disease recurrence or progression during/after first-line treatment including PD-(L)1 combined with chemotherapy, and PD-(L)1 monotherapy for advanced or metastatic disease.
6. Measurable disease by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Subjects are eligible if CNS metastases are asymptomatic or treated.
9. Life expectancy ≥12 weeks.
10. Fertile female must agree to use adequate contraception within 24 weeks from the beginning of the first dose of study medication to the last dose.
11. Adequate organ and marrow function.

Exclusion Criteria:

1. Prior treatment with anti-tumor virus, or prior T cell co-stimulation factors,including anti-Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody or other T cell-targeted drugs.
2. Subjects who had discontinued prior treatment due to immune-related adverse events (irAEs) or who are not suitable for PD-(L)1 treatment assessed by the investigator.
3. Subjects with histologically or cytologically-documented squamous cell NSCLC.
4. Prior treatments with anti-angiogenic agents.
5. Subjects with activated EGFR gene mutation or ALK fusion mutation.
6. Untreated or active central nervous system metastases (such as brain or meningeal metastases). Subjects are eligible if CNS metastases are asymptomatic or treated and subjects are off corticosteroids for at least 2 weeks prior to first dose of study therapy.
7. Radiotherapy for the chest and whole brain should be completed within 4 weeks before the first dose of study drug (palliative radiotherapy for bone lesions should be completed before the first dose of study drugs).
8. History of active or recent history of known or suspected autoimmune disease.
9. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, radiation pneumonitis requiring steroid therapy, or evidence of active pneumonitis with clinical symptoms.
10. History of active tuberculosis regardless of prior treatment.
11. Malignancies other than NSCLC within 5 years prior to first administration of drugs, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome, such as cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical resection.
12. Known mental illness, alcohol abuse, inability to quit smoking, drug or drug abuse, etc.
13. Active hepatitis B or hepatitis C; History of known HIV-positive history or known AIDS.
14. Treatment with any investigational agent within 28 days of signing ICF.
15. According to the judgment of the investigator, subjects have other factors that may cause the study to be terminated halfway, such as non-compliance with the protocol, other serious diseases (including mental illness) requiring combined treatment, severe laboratory abnormalities, and Factors such as family or society will affect the safety of subjects or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 1 year
  PFS is determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 1 year
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR:
  Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by investigator.
Duration of Response | up to 1 year
  Duration of Response, determined using RECIST v1.1 criteria
Disease Control Rate (DCR) | up to 1 year
  Disease Control Rate, determined using RECIST v1.1 criteria
Overall Survival (OS) | up to 2 years
  Overall survival is the time interval from the date of randomization to death due to any reason or lost of follow-up
Adverse Events (AEs) and Serious Adverse Events(SAEs) | up to 1 year
  The number of participants experiencing an AE and SAE will be assessed.Adverse
QLQ-LC13 | up to 1 years
  Quality of Life questionnaire lung cancer module 13
EORTCQLQ-C30 | up to 1 years
  European Organization for Reasearch and Treatment of Cancer C30

CONTACTS AND LOCATIONS:
Locations (1):
- China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xing P, Wang M, Zhao J, Zhong W, Chi Y, Xu Z, Li J. Study protocol: A single-arm, multicenter, phase II trial of camrelizumab plus apatinib for advanced nonsquamous NSCLC previously treated with first-line immunotherapy. Thorac Cancer. 2021 Oct;12(20):2825-2828. doi: 10.1111/1759-7714.14113. Epub 2021 Aug 18. PMID 34409776